CLINICAL TRIAL: NCT01278030
Title: Real Time 3-Dimensional Echocardiography for Left Ventricular Lead Site Selection to Reduce Cardiac Resynchronization Therapy Non-Responder Rates (ENVISION)
Brief Title: Real Time 3-Dimensional Echocardiography for Left Ventricular Lead Site Selection to Reduce Cardiac Resynchronization Therapy Non-Responder Rates
Acronym: ENVISION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRD 534
Record Dates: First submitted 2011-01-12; First posted 2011-01-17 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Patients will be implanted according to the standard of care with the LV lead in the traditional LV lead position.
- 3D echo-guided LV lead placement group (Experimental): Information about left ventricular mechanical dyssynchrony and the location of the site of latest mechanical activation based on Real-Time 3-Dimensional Echocardiography (RT3DE) will be available to the physician at the time of implant. This location will be used as the target for optimal LV lead placement.
  Interventions: Procedure: 3D echo-guided LV lead placement

INTERVENTIONS:
Procedure: 3D echo-guided LV lead placement — Information about left ventricular mechanical dyssynchrony and the location of the site of latest mechanical activation based on RT3DE will be available to the physician from the core lab analysis. This location will be used as the target for optimal LV lead placement.
  Arms: 3D echo-guided LV lead placement group

SUMMARY:
The purpose of this study is to demonstrate that cardiac resynchronization therapy (CRT) responder rate can be improved by 3-dimensional (3D) echo-guided left ventricular (LV) lead placement compared to traditional LV lead placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be implanted with an FDA approved St. Jude Medical CRT-D device (i.e. PROMOTE® or newer devices with similar functionality)
* Patients will have an approved indication per American College of Cardiology/American Heart Association/Heart Rhythm Society guidelines for implantation of a CRT-D
* Patients will receive a new implant or an upgrade from an existing pacemaker or Implantable Cardiovertor Defibrillator with no prior Left Ventricular lead placement
* Patients must be in sinus rhythm at the time of enrollment visit and baseline measurements

Exclusion Criteria:

* Persistent or permanent atrial fibrillation
* Heart transplantation
* Recent myocardial infarction (< 90 days)
* Contra-indication to contrast agent
* Are less than 18 years of age
* Are pregnant
* Are currently participating in a clinical investigation that includes an active treatment arm
* Have a life expectancy of less than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Heart Group, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 3D Echo-guided LV Lead Placement: The location of the site of latest mechanical activation based on 3-D Echo will be available to the physician from the core lab analysis. This location will be used as the target for optimal Left Ventricular lead placement.
- Control: Patients will be implanted according to the standard of care with the Left Ventricular lead in the traditional Left Ventricular lead position.
Period: Overall Study
Arm/Group | 3D Echo-guided LV Lead Placement | Control
Started | 43 | 35
Completed | 35 | 31
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3D Echo-guided LV Lead Placement | Control | Total
Number analyzed (Participants) | 43 | 35 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 13 | 31
  >=65 years | 25 | 22 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (13) | 67 (11) | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 28 | 26 | 54
Region of Enrollment [Number; unit: participants]
  United States | 43 | 35 | 78

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate
Description: The responder rate is defined as the proportion of patients with reduction in end systolic volume greater than or equal to 15%. The primary endpoint is the responder rate.
Time Frame: At 6 month follow-up
Population: Patients who completed the 6 month follow-up with implant 3D echo data.
Measure: Number; unit: percentage of participants
Arm/Group | 3D Echo-guided LV Lead Placement | Control
Number analyzed (Participants) | 33 | 25
percentage of participants | 67 | 60

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 3D Echo-guided LV Lead Placement | Control
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/35
Other Adverse Events (participants affected / at risk) | 1/43 | 1/35
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3D Echo-guided LV Lead Placement (N=43) | Control (N=35)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pericardial Effusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No